CLINICAL TRIAL: NCT03109769
Title: The Effect of Using Mobile Applications for Improving Oral Hygiene in Patients With Orthodontic Fixed Appliances: A Randomized Controlled Trial
Brief Title: The Effect of Using Mobile Applications for Improving Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Lecturer, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FUGRP/2014/191
Record Dates: First submitted 2017-04-05; First posted 2017-04-12 (Actual); Results first posted 2017-11-01 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone application (Experimental): Subjects in this group received a mobile phone application that sends active reminder notifications of oral hygiene 3 times a day.
  Interventions: Behavioral: Mobile phone application
- Verbal oral hygiene instructions (Active Comparator): Subjects in this group received verbal oral hygiene instructions during their regular orthodontic visits every 4 weeks.
  Interventions: Behavioral: Verbal oral hygiene instructions

INTERVENTIONS:
Behavioral: Mobile phone application
  Arms: Mobile phone application
Behavioral: Verbal oral hygiene instructions
  Arms: Verbal oral hygiene instructions

SUMMARY:
The study aims to investigate the effect of the use of mobile phone application sending reminders to patients with orthodontic fixed appliances on oral hygiene.

DETAILED DESCRIPTION:
Subjects were randomized into two groups, the first group received a mobile application that sends active reminders notifications of oral hygiene. The second group received verbal oral hygiene instructions during their regular visits to the orthodontics clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were having orthodontic fixed appliance treatment.
2. Participants were aged 12 years old and above, owned mobile phones and did not have mental or physical disabilities.
3. Participants were willing to comply with given oral hygiene instructions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar H AlKadhi, BDS, MS, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alkadhi OH, Zahid MN, Almanea RS, Althaqeb HK, Alharbi TH, Ajwa NM. The effect of using mobile applications for improving oral hygiene in patients with orthodontic fixed appliances: a randomised controlled trial. J Orthod. 2017 Sep;44(3):157-163. doi: 10.1080/14653125.2017.1346746. Epub 2017 Jul 13. PMID 28705122

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Phone Application: Subjects in this group received a mobile phone application that sends active reminder notifications of oral hygiene 3 times a day.
  Mobile phone application
- Verbal Oral Hygiene Instructions: Subjects in this group received verbal oral hygiene instructions during their regular orthodontic visits every 4 weeks.
  Verbal oral hygiene instructions
Period: Overall Study
Arm/Group | Mobile Phone Application | Verbal Oral Hygiene Instructions
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Phone Application | Verbal Oral Hygiene Instructions | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (3.2) | 17.2 (5.2) | 16.9 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 11 | 8 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Saudi Arabia | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Plaque Index
Description: Plaque index: 0, no plaque, 1, plaque seen on the tip of the explorer or with disclosing agent, 2. plaque seen with the naked eye, 3, abundance of plaque.
Time Frame: At baseline and after 4 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Phone Application | Verbal Oral Hygiene Instructions
Number analyzed (Participants) | 22 | 22
units on a scale
  Plaque index at baseline | 0.8050 (0.4062) | 0.8959 (0.4824)
  Plaque index after 4 weeks | 0.6677 (0.3146) | 0.9891 (0.5244)
Statistical Analysis 1: Comparison: Mobile Phone Application vs Verbal Oral Hygiene Instructions; The sample size was calculated as 44 participants. Sample size calculation was carried out through a pilot study on 30 participants with the group I mean=1.31, SD=0.39 and group II mean=1.62, SD=0.30, with ⍺=0.05 and 80% power. The null hypothesis was: there is no difference in plaque index and gingival index between verbal oral hygiene instructions and oral hygiene instructions using mobile applications in patients with orthodontic fixed appliances; Test type: Superiority; p = 0.0444, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Mobile Phone Application; Test type: Superiority; p = 0.0002, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.1373 — Difference in plaque index within the first group (mobile phone application) at 4 weeks compared to baseline. The mean difference was calculated as follows: plaque index at 4 weeks - plaque index at baseline
Statistical Analysis 3: Comparison: Mobile Phone Application; Test type: Superiority; p = 0.0283, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0932 — Difference in plaque index within the second group (verbal oral hygiene instructions) at 4 weeks compared to baseline. The mean difference was calculated as follows: plaque index at 4 weeks - plaque index at baseline

2. Primary Outcome: Change in Gingival Index
Description: Gingival index: 0, normal gingiva, 1, mild inflammation - slight change in color, slight edema and no bleeding on probing, 2, moderate inflammation - redness, edema and glazing and bleeding on probing, 3, severe inflammation - marked redness and edema, ulceration and tendency to spontaneous bleeding.
Time Frame: At baseline and after 4 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Phone Application | Verbal Oral Hygiene Instructions
Number analyzed (Participants) | 22 | 22
units on a scale
  Gingival index at baseline | 0.3450 (0.2955) | 0.4927 (0.3005)
  Gingival index after 4 weeks | 0.2273 (0.2256) | 0.5941 (0.5679)
Statistical Analysis 1: Comparison: Mobile Phone Application vs Verbal Oral Hygiene Instructions; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0283, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Mobile Phone Application; Test type: Superiority; p = 0.0002, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.1177 — Difference in gingival index within the first group (mobile phone application) at 4 weeks compared to baseline. The mean difference was calculated as follows: gingival index at 4 weeks - gingival index at baseline
Statistical Analysis 3: Comparison: Verbal Oral Hygiene Instructions; Test type: Superiority; p = 0.4809, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.1014 — Difference in gingival index within the second group (verbal oral hygiene instructions) at 4 weeks compared to baseline. The mean difference was calculated as follows: gingival index at 4 weeks - gingival index at baseline

ADVERSE EVENTS:
Arm/Group | Mobile Phone Application | Verbal Oral Hygiene Instructions
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No